CLINICAL TRIAL: NCT04774068
Title: A Phase I Study of Romidepsin in Combination With Parsaclisib in Relapsed and Refractory T-Cell Lymphomas
Brief Title: Romidepsin and Parsaclisib for the Treatment of Relapsed or Refractory T-Cell Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Walter Hanel (Other)
Responsible Party: Sponsor-Investigator, Walter Hanel, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-19264; NCI-2021-00728 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-02-19; First posted 2021-02-26 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Recurrent Anaplastic Large Cell Lymphoma; Recurrent Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Recurrent Transformed Mycosis Fungoides; Refractory Anaplastic Large Cell Lymphoma; Refractory Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Refractory Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Refractory Transformed Mycosis Fungoides; T-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell; Lymphoma, T-Cell, Cutaneous | interventions — parsaclisib; romidepsin; Depsipeptides; Lactones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (romidepsin, parsaclisib) (Experimental): PRE-PHASE: Patients receive romidepsin IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  INDUCTION PHASE: Patients receive romidepsin IV over 4 hours on days 1,8, and 15 and parsaclisib PO QD on days 1-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive romidepsin IV over 4 hours on days 1, 8, and 15 and parsaclisib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Parsaclisib; Drug: Romidepsin

INTERVENTIONS:
Drug: Parsaclisib — Given PO
  Other Names: (4R)-4-(3-((1S)-1-(4-Amino-3-methyl-1H-pyrazolo(3,4-d)pyrimidin-1-yl)ethyl)-5-chloro-2-ethoxy-6-fluorophenyl)pyrrolidin-2-one; INCB 50465; INCB-50465; INCB050465; INCB50465; WHO 10589
Drug: Romidepsin — Given IV
  Other Names: Antibiotic FR 901228; Depsipeptide; FK228; FR901228; Istodax; N-[(3S,4E)-3-Hydroxy-7-mercapto-1-oxo-4-heptenyl]-D-valyl-D-cysteinyl-(2Z)-2-amino-2-butenoyl-L-valine, (4->1) Lactone, Cyclic

SUMMARY:
This phase I trial finds the appropriate parsaclisib dose level in combination with romidepsin for the treatment of T-cell lymphomas that have come back (relapsed) or that have not responded to standard treatment (refractory). The other goals of this trial are to find the proportion of patients whose cancer is put into complete remission or significantly reduced by romidepsin and parsaclisib, and to measure the effectiveness of romidepsin and parsaclisib in terms of patient survival. Romidepsin blocks certain enzymes (histone deacetylases) and acts by stopping cancer cells from dividing. Parsaclisib is a PI3K inhibitor. The PI3K pathway promotes cancer cell proliferation, growth, and survival. Parsaclisib, thus, may stop the growth of cancer cells by blocking PI3K enzymes needed for cell growth. Giving romidepsin and parsaclisib in combination may work better in treating relapsed or refractory T-cell lymphomas compared to either drug alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) of parsaclisib in combination with romidepsin.

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR) of parsaclisib in combination with romidepsin in patients with relapsed/refractory primary cutaneous T-cell non-Hodgkin lymphoma / mature T-cell and NK-cell non-Hodgkin lymphoma (CTCL/PTCL).

II. To determine the duration of response (DOR) to treatment. III. Disease control rate (DCR). IV. To determine the progression-free survival (PFS) and overall survival (OS) of parsaclisib in combination with romidepsin in patients with relapsed/refractory CTCL/PTCL.

OUTLINE: This is a dose-escalation study of parsaclisib in the Induction Phase and fixed-dose in the Maintenance phase, and fixed-dose romidepsin in all Phases.

PRE-PHASE: Patients receive romidepsin intravenously (IV) over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

INDUCTION PHASE: Patients receive romidepsin IV over 4 hours on days 1,8, and 15 and parsaclisib orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE PHASE: Patients receive romidepsin IV over 4 hours on days 1, 8, and 15 and parsaclisib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Able to understand and voluntarily sign a consent form
* Biopsy proven diagnosis of PTCL or CTCL
* Relapsed/refractory PTCL, progressing after at least one line of systemic therapy (for anaplastic large cell lymphoma [ALCL], must have had prior treatment with brentuximab vedotin). OR
* Relapsed/Refractory CTCL, that progressed on at least 2 lines of skin-directed (topical) therapy and/or one line of systemic therapy. Pre-treatment with mogamulizumab and/or brentuximab vedotin (in the presence of CD30 positive disease) is NOT required as a criterion for eligibility. Skin-directed therapies include, but are not limited to topical steroids, topical chemotherapy, imiquimod, narrow band ultraviolet B (UVB), psoralen plus ultraviolet A photochemotherapy (PUVA), total skin electron beam radiation, and extracorporeal photopheresis
* Mycosis fungoides with large cell transformation is eligible
* Performance status (Eastern Cooperative Oncology Group [ECOG]) 0-2
* Life expectancy >= 90 days
* Patient must have at least stage IB CTCL (> 10% eBSA) or PTCL with disease defined by a nodal area of at least 1.5 cm in long dimension, extranodal disease of at least 1 cm in long dimension, or fludeoxyglucose F-18 - positron emission tomography (FDG-PET) avid disease (Deauville score = 5)
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 100,000/mm^3
* Calculated creatinine clearance >= 50mL/min (Cockcroft-Gault method)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal (ULN) or =< 5 x ULN if liver involved by lymphoma
* Bilirubin =< 2.0 x ULN. If the subject has Gilbert's disease, low-grade hemolysis, or liver involvement with lymphoma, a bilirubin level of =< 4 x ULN will be allowed
* Negative serum pregnancy test at the time of enrollment for females of childbearing potential
* Women of childbearing potential (as defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal for at least 24 consecutive months) are required to use a highly effective method of contraception (i.e. intrauterine device [IUD], hormonal [birth control pills, injections, or implants] while on study). Male patients engaged in a sexual relationship with a woman of childbearing potential must agree to use a latex condom during sexual contact, even if he has had a successful vasectomy
* All cancer therapy, including radiation, topical steroid, and chemotherapy must have been discontinued at least 1 week or 3 half-lives whichever is the longest prior to treatment in this study. The only exceptions are participants who are symptomatic from their skin lesions and have been on corticosteroids for prolonged periods of time (> 60 days) without change may continue use of either systemic steroids (equivalent to < 10 mg per day of prednisone) or topical steroids are eligible for this study if the frequency and dosage steroids has not changed for 14 days prior to the study

Exclusion Criteria:

* Patients with uncontrolled central nervous system (CNS) disease
* Use of immunosuppressive therapy within 28 days of randomization. Immunosuppressive therapy includes, but is not limited to, cyclosporine A, tacrolimus, or high-dose corticosteroids. Participants receiving corticosteroids must be at a dose of =< 10 mg/day prednisone (or equivalent) within 7 days of randomization. However, topical steroids (maximum strength Class III according to World Health Organization Classification of Topical steroids) are allowed to control pruritis
* An active infection requiring a systemic antimicrobial. The patient should be off antibiotic treatment for an active infection for 7 days prior to enrollment in the trial. However, antibiotic prophylaxis is acceptable as long as the dose of the medication has been stable for at least 7 days prior to the baseline exam
* Exposure to a live vaccine within 30 days of treatment start
* Positive at the time of screening for human immunodeficiency virus (HIV), hepatitis B surface antigen or viral load, hepatitis C viral load. Hepatitis B (HBV) or hepatitis C (HCV) infection: Participants positive for HBV surface antigen or HBV core antibody will be eligible if they are negative for HBV-deoxyribonucleic acid (DNA); these participants should be considered for prophylactic antiviral therapy. Participants positive for anti-HCV antibody will be eligible if they are negative for HCV ribonucleic acid (RNA)
* Prior malignancy within the past 2 years (allowing squamous cell and basal cell carcinomas with free margins at excision)
* Prior treatment with a PI3K inhibitor
* Presence of an abnormal electrocardiogram (ECG) that is clinically meaningful. Screening corrected QT interval (QTc) interval > 450 milliseconds is excluded (corrected by Fridericia). In the event that a single QTc is > 450 milliseconds, the participant may enroll if the average QTc for 3 ECGs is < 450 milliseconds. If left bundle branch is present, upper limit of QTc will be 550 milliseconds
* Use of strong CYP3A4 inhibitors and inducers. If a CYP3A4 inhibitor was recently used, there should be 14 days or 5 half-lives time (whichever is longer) before the first dose of parsaclisib is administered. Use of moderate CYP3A4 inhibitors are strongly discouraged but not strictly prohibited. If a strong CYP3A4 inhibitor is started after study enrollment, the study principal investigator (PI) should be contacted to discuss alternatives
* Unable to swallow tablets, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction likely to interfere with the delivery, absorption, or metabolism of parsaclisib
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Progression while on romidepsin or within 3 months of discontinuation of romidepsin. Prior treatment with romidepsin is allowed if it was well-tolerated
* Unwillingness to comply with study procedures, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the investigator
* Pregnant or lactating, or intending to become pregnant during the study
* Clinically significant abnormalities in medical history, physical examination, or laboratory values, which in the opinion of the investigator would make the patient unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of parsaclisib | Cycles 3-5 (each cycle is 28 days)
  Will use a time-to-event Bayesian optimal interval design to identify the MTD of this combination regimen.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 24 weeks
  ORR defined as the proportion of patients who achieve a complete or partial response among all evaluable patients. The proportion will be provided with a 95% binomial confidence interval. For mature T-Cell and NK-Cell Non-Hodgkin lymphoma (PTCL) patients, response will be evaluated by the Lugano criteria. For primary cutaneous T-Cell Non-Hodgkin lymphoma (CTCL) patients, responses will be evaluated using the Global Response Score. ORR lasting >= 4 months will be captured for CTCL patients.
Duration of response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  DOR defined by time to progression; time from the first romidepsin dose until disease progression.
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS will be calculated from the start of the combination treatment to the time of progression or death, whichever occurs first. Will use the method of Kaplan-Meier to describe these survival endpoints; reporting median or estimates at certain time points with 95% confidence intervals.
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Will use the method of Kaplan-Meier to describe these survival endpoints; reporting median or estimates at certain time points with 95% confidence intervals.
Disease control rate (DCR) | Up to 2 years
  DCR is defined as the proportion of patients with complete response, partial response, or stable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Hanel, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT04774068/ICF_000.pdf